CLINICAL TRIAL: NCT03162159
Title: An Adult Height Prediction Model for Congenital Adrenal Hyperplasia From a National Cohort (OPALE Model Study)
Brief Title: Adult Height Prediction in Congenital Adrenal Hyperplasia
Acronym: OPALE Model
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CE-CIC-GREN-09-19
Record Dates: First submitted 2017-05-11; First posted 2017-05-22 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cohort for model computing: patients with CAH, born between 1970 and 1993, with genetically proven CAH, available growth and bone maturation data.
  Interventions: Other: Collection of growth and bone maturation data
- cohort for model validation: patients with CAH, born between 1994 and 1998, with genetically proven CAH, available growth and bone maturation data.
  Interventions: Other: Collection of growth and bone maturation data

INTERVENTIONS:
Other: Collection of growth and bone maturation data

SUMMARY:
Congenital Adrenal Hyperplasia (CAH) is a genetic rare disease, which alters the adrenal production of gluco and mineralo corticoïds. The treatment consists in supplementing children with hydrocortisone. Despite care for these children has improved substantially across decades, short adult height (AH) still remains an important consequence of the disease. About 20% of patients have an AH below 2 standard deviations compared to their expected AH.

In the OPALE-Model study, the investigators want to collect data from a cohort of 496 CAH French patients, born between 1970 and 1991 with a known genotype. Using their age, sex, growth, disease, bone maturation and pubertal data, the investigators will build a model which allows to predict their AH using data available at 8 years of age. The growth charts built from this cohort have shown that currently used formula to calculate the predicted AH (Bayley-Pineau's formula) is not applicable to children with CAH.

In this project, the investigators plan to compute an AH prediction model using data from children born between 1970 and 1993, and to validate the model using data from a different cohort (i.e. children born between 1994 and 1998). this choice was due to availability of data for computing the model first, and in a second stage, data from more recently born patients.

ELIGIBILITY:
Inclusion Criteria:

* children with CAH, genetically proven, classical form, virilizing form, with deficit of 21 hydroxylase, 11 beta hydroxylase, or 3 beta ol dehydrogenase, born between 1972-1993 (cohort 1) and 1994-1998 (cohort 2).
* medical charts should be available.

Exclusion Criteria:

* Patients with chronic growth altering disease, Turner syndrome, or other genetic anomaly
* Patients having received any treatment with Growth Hormone (GH)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adullts with Congenital Adrenal Hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 496 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Adult height (AH) | up to 18 years
  AH is defined as i) the height recorded after age 20 in boys or 18 in girls; ii) Or the height recorded when bone age is >= 18 years in boys and 16 years in girls; Or iii) the height measured after growth velocity dropped to <= 1 cm/year.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Cornu, MD, Study Chair — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bretones P, Riche B, Pichot E, David M, Roy P, Tardy V, Kassai B, Gaillard S, Bernoux D, Morel Y, Chatelain P, Nicolino M, Cornu C; French Collaborative CAH Growth Study Group. Growth curves for congenital adrenal hyperplasia from a national retrospective cohort. J Pediatr Endocrinol Metab. 2016 Dec 1;29(12):1379-1388. doi: 10.1515/jpem-2016-0156. PMID 27852974